CLINICAL TRIAL: NCT06489379
Title: High Flow Nasal Oxygen for Acute Hypoxemic Respiratory Failure in the Emergency Room: the GLAMOUR Study
Brief Title: High Flow Nasal Oxygen for Acute Hypoxemic Respiratory Failure in the Emergency Room
Acronym: GLAMOUR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, FRANCESCHI FRANCESCO, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6697
Record Dates: First submitted 2024-06-21; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Respiratory Distress Syndrome, Adult
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- standard oxygen (Active Comparator)
  Interventions: Other: standard oxygen
- high flow nasal oxygen (Experimental)
  Interventions: Device: high flow nasal cannula

INTERVENTIONS:
Device: high flow nasal cannula — humidified and heated oxygen
  Arms: high flow nasal oxygen
Other: standard oxygen — oxygen delivery through Venturi mask
  Arms: standard oxygen

SUMMARY:
The aim of this multicenter, randomized, controlled, open-label trial is to investigate the efficacy of early treatment with HFNO compared with SOT in preventing early deterioration of patients admitted to the ER because of acute hypoxemic respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* PaO2/FiO2 ratio between 250 and 150 mmHg or SpO2/FiO2 ratio between 190 and 274, after at least 15 minutes of spontaneous breathing through a Venturi mask (VM), with a FiO2 targeted at a SpO2 94-97%;
* Respiratory rate(RR)≤35breaths/min,afteratleast15minutesofspontaneous breathing through a VM, with a FiO2 targeted at a SpO2 94-97%;
* PaCO2 ≤ 45 mmHg;
* Unilateral or bilateral infiltrate(s), as detected with chest radiography and/or computed tomography and/or with lung ultrasound not fully explained by effusions, atelectasis, or nodules/masses. Infiltrates at lung ultrasound are defined as presence of focal B-lines, consolidations (with irregular marginal contour, air bronchogram, air trapping sign) and irregularity of the pleural line.

Exclusion Criteria:

* Respiratory failure due to:

  * Acute asthma or COPD exacerbation,
  * Cardiac failure or fluid overload as primary cause of respiratory failure;
* Unstable angina or ongoing acute myocardial infarction;
* Acute respiratory acidosis with pH < 7.35 and PaCO2 > 45 mmHg;
* Hemodynamic instability and/or use of vasopressors/inotropes;
* Altered mental status (Kelly >3), see Figure 1;(18)
* Contraindications to NIV (high risk of aspiration pneumonia, impaired airways protection, head-facial trauma and/or burns, uncooperative patient, cranial/thoracic/abdominal open wounds);
* Indications to urgent intubation performed according to the clinician in charge;
* Body Mass Index > 35 kg/m2;
* Pregnancy;
* Patient's refusal to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Early deterioration | 24 hours
  occurrence of any of the following from randomization: respiratory worsening; respiratory acidosis; severe respiratory distress; start of non-invasive ventilation; necessity of endotracheal intubation; development of shock; death.

SECONDARY OUTCOMES:
Development of respiratory acidosis | 2, 12 and 24 hours
  arterial pH
Development of hypercapnia | 2, 12 and 24 hours
  arterial pCO2
Worsening hypoxemia | 2, 12 and 24 hours
  P/F ratio
Worsening respiratory distress | 2, 12 and 24 hours
  respiratory frequency
duration of any type of ventilatory support | 90 days
  hours of ventilatory support
rate of ICU admission | 90 days
  number of patients admitted to ICU
hospital length-of-stay | 30 days
  duration of hospitalization
in-hospital mortality | 90 days
  death during hospitalization
ICU length-of-stay | 90 days
  duration of ICU stay
ICU mortality | 90 days
  death in ICU
development of complications | 90 days
  composite outcome of septic shock, nosocomial pneumonia, cardiac arrhythmia, cardiac arrest, delirium
level of dyspnea | 24 hours
  utilizing Borg scale
patient comfort | 24 hours
  utilizing visual analogue scale
clinical setting after ED stabilization | 24 hours
  type of ward admission
standard vs asymmetrical high-flow nasal cannula | 24 hours
  rate of early deterioration in the treatment group will be compared between patients treated with standard or asymmetrical high-flow nasal cannula

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Raveling T, Vonk J, Struik FM, Goldstein R, Kerstjens HA, Wijkstra PJ, Duiverman ML. Chronic non-invasive ventilation for chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2021 Aug 9;8(8):CD002878. doi: 10.1002/14651858.CD002878.pub3. PMID 34368950
- [Background] Berbenetz N, Wang Y, Brown J, Godfrey C, Ahmad M, Vital FM, Lambiase P, Banerjee A, Bakhai A, Chong M. Non-invasive positive pressure ventilation (CPAP or bilevel NPPV) for cardiogenic pulmonary oedema. Cochrane Database Syst Rev. 2019 Apr 5;4(4):CD005351. doi: 10.1002/14651858.CD005351.pub4. PMID 30950507
- [Background] Rochwerg B, Brochard L, Elliott MW, Hess D, Hill NS, Nava S, Navalesi P Members Of The Steering Committee, Antonelli M, Brozek J, Conti G, Ferrer M, Guntupalli K, Jaber S, Keenan S, Mancebo J, Mehta S, Raoof S Members Of The Task Force. Official ERS/ATS clinical practice guidelines: noninvasive ventilation for acute respiratory failure. Eur Respir J. 2017 Aug 31;50(2):1602426. doi: 10.1183/13993003.02426-2016. Print 2017 Aug. PMID 28860265
- [Background] Antonelli M, Conti G, Esquinas A, Montini L, Maggiore SM, Bello G, Rocco M, Maviglia R, Pennisi MA, Gonzalez-Diaz G, Meduri GU. A multiple-center survey on the use in clinical practice of noninvasive ventilation as a first-line intervention for acute respiratory distress syndrome. Crit Care Med. 2007 Jan;35(1):18-25. doi: 10.1097/01.CCM.0000251821.44259.F3. PMID 17133177
- [Background] Carteaux G, Millan-Guilarte T, De Prost N, Razazi K, Abid S, Thille AW, Schortgen F, Brochard L, Brun-Buisson C, Mekontso Dessap A. Failure of Noninvasive Ventilation for De Novo Acute Hypoxemic Respiratory Failure: Role of Tidal Volume. Crit Care Med. 2016 Feb;44(2):282-90. doi: 10.1097/CCM.0000000000001379. PMID 26584191
- [Background] Bellani G, Laffey JG, Pham T, Madotto F, Fan E, Brochard L, Esteban A, Gattinoni L, Bumbasirevic V, Piquilloud L, van Haren F, Larsson A, McAuley DF, Bauer PR, Arabi YM, Ranieri M, Antonelli M, Rubenfeld GD, Thompson BT, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators; ESICM Trials Group. Noninvasive Ventilation of Patients with Acute Respiratory Distress Syndrome. Insights from the LUNG SAFE Study. Am J Respir Crit Care Med. 2017 Jan 1;195(1):67-77. doi: 10.1164/rccm.201606-1306OC. PMID 27753501
- [Background] Demoule A, Girou E, Richard JC, Taille S, Brochard L. Benefits and risks of success or failure of noninvasive ventilation. Intensive Care Med. 2006 Nov;32(11):1756-65. doi: 10.1007/s00134-006-0324-1. Epub 2006 Sep 21. PMID 17019559
- [Background] Marjanovic N, Guenezan J, Frat JP, Mimoz O, Thille AW. High-flow nasal cannula oxygen therapy in acute respiratory failure at Emergency Departments: A systematic review. Am J Emerg Med. 2020 Jul;38(7):1508-1514. doi: 10.1016/j.ajem.2020.04.091. Epub 2020 May 4. PMID 32389397
- [Background] Roca O, Riera J, Torres F, Masclans JR. High-flow oxygen therapy in acute respiratory failure. Respir Care. 2010 Apr;55(4):408-13. PMID 20406507
- [Background] Oczkowski S, Ergan B, Bos L, Chatwin M, Ferrer M, Gregoretti C, Heunks L, Frat JP, Longhini F, Nava S, Navalesi P, Ozsancak Ugurlu A, Pisani L, Renda T, Thille AW, Winck JC, Windisch W, Tonia T, Boyd J, Sotgiu G, Scala R. ERS clinical practice guidelines: high-flow nasal cannula in acute respiratory failure. Eur Respir J. 2022 Apr 14;59(4):2101574. doi: 10.1183/13993003.01574-2021. Print 2022 Apr. PMID 34649974
- [Background] Chidekel A, Zhu Y, Wang J, Mosko JJ, Rodriguez E, Shaffer TH. The effects of gas humidification with high-flow nasal cannula on cultured human airway epithelial cells. Pulm Med. 2012;2012:380686. doi: 10.1155/2012/380686. Epub 2012 Sep 3. PMID 22988501
- [Background] Frat JP, Thille AW, Mercat A, Girault C, Ragot S, Perbet S, Prat G, Boulain T, Morawiec E, Cottereau A, Devaquet J, Nseir S, Razazi K, Mira JP, Argaud L, Chakarian JC, Ricard JD, Wittebole X, Chevalier S, Herbland A, Fartoukh M, Constantin JM, Tonnelier JM, Pierrot M, Mathonnet A, Beduneau G, Deletage-Metreau C, Richard JC, Brochard L, Robert R; FLORALI Study Group; REVA Network. High-flow oxygen through nasal cannula in acute hypoxemic respiratory failure. N Engl J Med. 2015 Jun 4;372(23):2185-96. doi: 10.1056/NEJMoa1503326. Epub 2015 May 17. PMID 25981908
- [Background] Tinelli V, Cabrini L, Fominskiy E, Franchini S, Ferrante L, Ball L, Pelosi P, Landoni G, Zangrillo A, Secchi A. High Flow Nasal Cannula Oxygen vs. Conventional Oxygen Therapy and Noninvasive Ventilation in Emergency Department Patients: A Systematic Review and Meta-Analysis. J Emerg Med. 2019 Sep;57(3):322-328. doi: 10.1016/j.jemermed.2019.06.033. Epub 2019 Aug 14. PMID 31421952
- [Background] Rochwerg B, Granton D, Wang DX, Helviz Y, Einav S, Frat JP, Mekontso-Dessap A, Schreiber A, Azoulay E, Mercat A, Demoule A, Lemiale V, Pesenti A, Riviello ED, Mauri T, Mancebo J, Brochard L, Burns K. High flow nasal cannula compared with conventional oxygen therapy for acute hypoxemic respiratory failure: a systematic review and meta-analysis. Intensive Care Med. 2019 May;45(5):563-572. doi: 10.1007/s00134-019-05590-5. Epub 2019 Mar 19. PMID 30888444
- [Background] Matthay MA, Arabi Y, Arroliga AC, Bernard G, Bersten AD, Brochard LJ, Calfee CS, Combes A, Daniel BM, Ferguson ND, Gong MN, Gotts JE, Herridge MS, Laffey JG, Liu KD, Machado FR, Martin TR, McAuley DF, Mercat A, Moss M, Mularski RA, Pesenti A, Qiu H, Ramakrishnan N, Ranieri VM, Riviello ED, Rubin E, Slutsky AS, Thompson BT, Twagirumugabe T, Ware LB, Wick KD. A New Global Definition of Acute Respiratory Distress Syndrome. Am J Respir Crit Care Med. 2024 Jan 1;209(1):37-47. doi: 10.1164/rccm.202303-0558WS. PMID 37487152
- [Background] Rice TW, Wheeler AP, Bernard GR, Hayden DL, Schoenfeld DA, Ware LB; National Institutes of Health, National Heart, Lung, and Blood Institute ARDS Network. Comparison of the SpO2/FIO2 ratio and the PaO2/FIO2 ratio in patients with acute lung injury or ARDS. Chest. 2007 Aug;132(2):410-7. doi: 10.1378/chest.07-0617. Epub 2007 Jun 15. PMID 17573487
- [Background] Demi L, Wolfram F, Klersy C, De Silvestri A, Ferretti VV, Muller M, Miller D, Feletti F, Welnicki M, Buda N, Skoczylas A, Pomiecko A, Damjanovic D, Olszewski R, Kirkpatrick AW, Breitkreutz R, Mathis G, Soldati G, Smargiassi A, Inchingolo R, Perrone T. New International Guidelines and Consensus on the Use of Lung Ultrasound. J Ultrasound Med. 2023 Feb;42(2):309-344. doi: 10.1002/jum.16088. Epub 2022 Aug 22. PMID 35993596
- [Background] Kelly BJ, Matthay MA. Prevalence and severity of neurologic dysfunction in critically ill patients. Influence on need for continued mechanical ventilation. Chest. 1993 Dec;104(6):1818-24. doi: 10.1378/chest.104.6.1818. PMID 8252971
- [Background] O'Driscoll BR, Howard LS, Earis J, Mak V. British Thoracic Society Guideline for oxygen use in adults in healthcare and emergency settings. BMJ Open Respir Res. 2017 May 15;4(1):e000170. doi: 10.1136/bmjresp-2016-000170. eCollection 2017. No abstract available. PMID 28883921
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Crimi C, Noto A, Madotto F, Ippolito M, Nolasco S, Campisi R, De Vuono S, Fiorentino G, Pantazopoulos I, Chalkias A, Libra A, Mattei A, Scala R, Clini EM, Ergan B, Lujan M, Winck JC, Giarratano A, Carlucci A, Gregoretti C, Groff P, Cortegiani A; COVID-HIGH Investigators. High-flow nasal oxygen versus conventional oxygen therapy in patients with COVID-19 pneumonia and mild hypoxaemia: a randomised controlled trial. Thorax. 2023 Apr;78(4):354-361. doi: 10.1136/thoraxjnl-2022-218806. Epub 2022 May 17. PMID 35580898
- [Background] Torres A, Sibila O, Ferrer M, Polverino E, Menendez R, Mensa J, Gabarrus A, Sellares J, Restrepo MI, Anzueto A, Niederman MS, Agusti C. Effect of corticosteroids on treatment failure among hospitalized patients with severe community-acquired pneumonia and high inflammatory response: a randomized clinical trial. JAMA. 2015 Feb 17;313(7):677-86. doi: 10.1001/jama.2015.88. PMID 25688779
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] Puntillo KA, White C, Morris AB, Perdue ST, Stanik-Hutt J, Thompson CL, Wild LR. Patients' perceptions and responses to procedural pain: results from Thunder Project II. Am J Crit Care. 2001 Jul;10(4):238-51. PMID 11432212
- [Background] Le Gall JR, Lemeshow S, Saulnier F. A new Simplified Acute Physiology Score (SAPS II) based on a European/North American multicenter study. JAMA. 1993 Dec 22-29;270(24):2957-63. doi: 10.1001/jama.270.24.2957. PMID 8254858
- [Background] Vincent JL, Moreno R, Takala J, Willatts S, De Mendonca A, Bruining H, Reinhart CK, Suter PM, Thijs LG. The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. On behalf of the Working Group on Sepsis-Related Problems of the European Society of Intensive Care Medicine. Intensive Care Med. 1996 Jul;22(7):707-10. doi: 10.1007/BF01709751. No abstract available. PMID 8844239